CLINICAL TRIAL: NCT01227031
Title: Pharmacogenomic Study of Androgenetic Alopecia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Taipei Medical University-Wan Fang Hospital, Department of Dermatology, Taipei Medical University-Wan Fang Hospital
Other Study IDs: 98089
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2010-11-12 (Estimated); Status verified 2010-10

CONDITIONS: Androgenetic Alopecia
Keywords: Genetic susceptibility of androgenetic alopecia; Genetic difference in Finasteride response
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extraction from blood sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Androgenic alopecia, the common form of hair loss is a highly heritable disorder of considerable social significance affecting around 40% of adult men and women. A variety of genetic and environmental factors are likely to play a role in androgenetic alopecia. Genetic variants in the human androgen receptor gene (AR) have been reported to be associated with AGA in Caucasians. Other genes involved with hair loss also have been found. One of them being a gene on chromosome 3 (3q26). A recent genome-wide association study in 296 individuals with male-pattern baldness and 347 controls had carried out and five SNPs on chromosome 20p11 were found to be highly significant association for AGA (rs2180439 combined P = 2.7 x 10(-15)). No interaction was detected with the X-chromosomal androgen receptor locus, suggesting that the 20p11 locus has a role in a yet-to-be-identified androgen-independent pathway.

The total number of evaluated patients with androgenic alopecia will be at least 300. All patients will be further grouped as good responders or poor responders to conventional medications, such as topical minoxidil and systemic finasteride. Candidate genes potentially involved in gout and its treatment response will be selected from the published literatures; specifically, two resources of candidate genes will be selected: (i) genes which are known to directly link with androgenic alopecia, and (ii) genes are potentially implicated in particular pathways of androgen/estrogen receptors, metabolism and downstream signals, and genes involved in anti-oxidants or hair growth. The SNP genotyping will be performed by MALDI-TOF Mass Spectrometry. Data analysis will be performed by comparing SNPs allele frequency between good responder and poor responder to conventional medications of patients with androgenic alopecia and further comparing to the allele frequency of SNPs in healthy controls. A functional study will also be done to prove the genetic association.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign inform consent form
* Willing to received history taking by telephone or interview
* Diagnosed androgenetic alopecia by Hamilton-Norwood classification
* More than 20 year-old, both sex

Exclusion Criteria:

* Ever had trauma over alopecia area
* Cancer, infection, or other systemic disease that might interfere diagnosis
* Unconfirmed diagnosis clinically or pathologically.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Androgenetic alopecia (pattern hair loss)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ren-Yu Tsai, Principal Investigator — Taipei Medical University-Wan Fang Hospital
Locations (1):
- Taipei Medical University-Wan Fang Hospital, Taipei, Taiwan